CLINICAL TRIAL: NCT04557943
Title: The Level of Cartilage Oligomeric Matrix Protein (COMP) and Urinary C-Terminal Telopeptides of Type II Collagen (uCTX-II) After Prolotherapy Intervention and The Functional Outcome in Patient With Knee Osteoarthritis
Brief Title: Prolotherapy Intervention Effect in Patient With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Researcher, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2708201904
Record Dates: First submitted 2020-09-07; First posted 2020-09-22 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; COMP; uCTX-II; Prolotherapy; Functional Outcome
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Prolotherapy; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: This study involves two arms assigned randomly for receiving different treatment. One arm for Prolotherapy and Sodium Hyaluronate in the comparison group.
Who Masked: Participant, Outcomes Assessor
Masking Description: A sealed envelope of the randomized sequence was given to the investigator and care provider, and participants were recruited consecutively according to the sequence. Participants were masked from the therapy by receiving treatment individually in different rooms and occasions. On the day of the assessment, the physician and laboratory technicians were blinded from group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Hyaluronate (Active Comparator): Hyaluronate sodium injection is performed intra-articularly using 2 mL of Adant® Disposable. The treatment will be given five times, on day 1st, 8th, 15th, 22nd, and 29th
  Interventions: Drug: Sodium Hyaluronate
- Prolotherapy (Experimental): Prolotherapy injection is performed intra-articularly and extra-articularly by a physician. Intra-articular injection with 25% dextrose will be carried out with the following details: 5 mL of 40% dextrose, 2 mL of lidocaine, and 1 mL of aqua dest are inserted into the 10-mL syringe, then 5 mL are injected with the superolateral approach. An extra-articular injection with 15% dextrose will be carried out with the following details:
  in the 10-mL syringe 4 mL of 40% dextrose, 2 mL lidocaine, and 4 mL of distilled water are injected, to make a total of 30-40 mL injections. Treatment will be carried out on day 1st, 29th, and 57th.
  Interventions: Drug: Prolotherapy

INTERVENTIONS:
Drug: Prolotherapy — Prolotherapy injection is performed intra-articularly and extra-articularly by a physician. Intra-articular injection with 25% dextrose will be carried out with the following details: 5 mL of 40% dextrose, 2 mL of lidocaine, and 1 mL of aqua dest are inserted into the 10-mL syringe, then 5 mL are injected with the superolateral approach. An extra-articular injection with 15% dextrose will be carried out with the following details:
  in the 10-mL syringe 4 mL of 40% dextrose, 2 mL lidocaine, and 4 mL of distilled water are injected, to make a total of 30-40 mL injections. Treatment will be carried out on day 1st, 29th, and 57th.
  Other Names: Prolotherapy Dextrose
  Arms: Prolotherapy
Drug: Sodium Hyaluronate — Hyaluronan sodium injection is performed intra-articularly using 2 mL of Adant® Disposable. The treatment will be given five times, on day 1st, 8th, 15th, 22nd, and 29th
  Other Names: 2 mL Sodium Hyaluronate
  Arms: Sodium Hyaluronate

SUMMARY:
Introduction :

Prolotherapy is regenerative tissue therapy which is considered to be efficacious in reducing symptoms and morbidity of Knee Osteoarthritis (KOA), but only a few studies demonstrate the effect of prolotherapy at the biomolecular level, particularly the level of Cartilage Oligomeric Matrix Protein (COMP), and Urinary C-Terminal Telopeptides of Type II Collagen (uCTX-II) as the biomarkers of cartilage repair.

Objective:

To determine the effect of prolotherapy on COMP and uCTX-II levels, and functional outcomes in KOA patients.

Method:

a double-blind randomized controlled trial study involving 36 participants who had been diagnosed with KOA. History taking, functional outcome assessment, COMP, and uCTX-II were measured. The prolotherapy via intraarticular and extraarticular was performed at Day-1, Day-29, and Day-57 followed by the evaluation of functional outcome, COMP, and uCTX-II at day 78

Alternative Hypothesis :

Prolotherapy provides improvement of cartilage based on COMP and UCTX-II levels and functional outcome among KOA patients

DETAILED DESCRIPTION:
Design :

Double-blind randomized trial

Randomization :

Simple Randomization generated by an online randomizer

Sample Size :

Difference between two means of primary outcome where

1. mean difference (μ 1 - μ 2 ) = 0.05
2. pool variance = 0.09
3. Z 1-α/2 = 1.95 with type 1 error 5%
4. 1-β = 1.282 with power 90%. Yielding 16 patients for each arm

Time Period of Recruitment September 2019- August 2020

Detailed Intervention

1. Intervention group : Prolotherapy given three times (Day-1, Day-29, and Day-57 )
2. Comparison group : Hyaluronate given five times (Day-1, Day-8, Day-15, Day-22, and Day-29.)

Outcome Measurement :

1. Cartilage Oligomeric Matrix Protein (COMP) Source of Sample : Median Cubital Vein Whole Blood Measurement : Enzyme-linked Immunoassay
2. Urinary C-Terminal Telopeptides of Type II Collagen (uCTX-II) Source of Sample : 50 cc of random urine sample Measurement : Enzyme-linked Immunoassay
3. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for functional Outcome (self-reported assessment)

Domains :

1. five elements of pain (score range 0-20),
2. two for stiffness (score range 0-8),
3. 17 for functional limitation (score range 0-68)

Classification :

0 - 24 : Mild 25 - 48 : Moderate 49 - 72 : Severe 73 - 96 : Extremely Severe

Statistical analysis :

1. Descriptive statistic to elaborate baseline characteristic
2. Assuming the baseline characteristic between groups are similar, the independent t-test will be conducted to see the differences between group, whereas Mann Whitney will be performed for non parametric data
3. Difference within group (baseline and last day) will be measured by paired-t test or wilcoxon for non parametric scenario

ELIGIBILITY:
Inclusion Criteria:

1. The patient provides consent to be part of the research.
2. The diagnosis of Knee Osteoarthritis was made based on clinical criteria/radiology American College of Rheumatology (ACR) 2012 with radiology grading according to Kellgren-Lawrence 2-3

Exclusion Criteria:

1. The Patient has received other forms of intraarticular injection therapy.
2. The patient has received Non Steroid Anti inflammation drug (NSAID) therapy for one week before the start of the intervention.
3. The patient has one or more contraindications for prolotherapy (e.g., Abscess, cellulitis, or septic arthritis).

Drop Out Criteria :

1. The patient has undergone a strenuous physical activity that precipitates a degree of complication (i.e., joint effusion).
2. The use of NSAID within one week after the intervention.
3. The patient does not adhere to the intervention.
4. The patient developed or being diagnosed with osteoarthritis or other forms of inflammatory disease in other joints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Cartilage Oligomeric Matrix Protein (COMP) | Measured on the first day before intervention and day 78 after the first dose of treatment in all groups
  cartilage oligomeric matrix protein from whole blood measured using Enzyme-linked Immunoassay (ELISA). Mean difference between group will be assessed

SECONDARY OUTCOMES:
Urinary C-Terminal Telopeptides of Type II Collagen (uCTX-II) | Measured on the first day before intervention and day 78 after the first injection on the prolotherapy group and Day 50 after the first injection for the hyaluronate group
  Urinary C-Terminal Telopeptides of Type II Collagen from urine sample measured using Enzyme-linked Immunoassay (ELISA)
Functional Outcome | Measured on the first day before intervention and day 78 after the first injection on the prolotherapy group and Day 50 after the first injection for the hyaluronate group
  the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index ) measuring three domains (pain, function limitation and stiffness) ranging from 0-96 of total score.

CONTACTS AND LOCATIONS:
Overall Officials: Yose Waluyo, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University, Faculty of Medicine, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rabago D, Zgierska A, Fortney L, Kijowski R, Mundt M, Ryan M, Grettie J, Patterson JJ. Hypertonic dextrose injections (prolotherapy) for knee osteoarthritis: results of a single-arm uncontrolled study with 1-year follow-up. J Altern Complement Med. 2012 Apr;18(4):408-14. doi: 10.1089/acm.2011.0030. PMID 22515800
- [Background] Eslamian F, Amouzandeh B. Therapeutic effects of prolotherapy with intra-articular dextrose injection in patients with moderate knee osteoarthritis: a single-arm study with 6 months follow up. Ther Adv Musculoskelet Dis. 2015 Apr;7(2):35-44. doi: 10.1177/1759720X14566618. PMID 25829954
- [Background] Rabago D, Patterson JJ, Mundt M, Kijowski R, Grettie J, Segal NA, Zgierska A. Dextrose prolotherapy for knee osteoarthritis: a randomized controlled trial. Ann Fam Med. 2013 May-Jun;11(3):229-37. doi: 10.1370/afm.1504. PMID 23690322
- [Background] Arias-Vazquez PI, Tovilla-Zarate CA, Legorreta-Ramirez BG, Burad Fonz W, Magana-Ricardez D, Gonzalez-Castro TB, Juarez-Rojop IE, Lopez-Narvaez ML. Prolotherapy for knee osteoarthritis using hypertonic dextrose vs other interventional treatments: systematic review of clinical trials. Adv Rheumatol. 2019 Aug 19;59(1):39. doi: 10.1186/s42358-019-0083-7. PMID 31426856
- [Background] Scarpellini M, Lurati A, Vignati G, Marrazza MG, Telese F, Re K, Bellistri A. Biomarkers, type II collagen, glucosamine and chondroitin sulfate in osteoarthritis follow-up: the "Magenta osteoarthritis study". J Orthop Traumatol. 2008 Jun;9(2):81-7. doi: 10.1007/s10195-008-0007-5. Epub 2008 May 28. PMID 19384621
- [Background] Garnero P, Conrozier T, Christgau S, Mathieu P, Delmas PD, Vignon E. Urinary type II collagen C-telopeptide levels are increased in patients with rapidly destructive hip osteoarthritis. Ann Rheum Dis. 2003 Oct;62(10):939-43. doi: 10.1136/ard.62.10.939. PMID 12972471
- [Background] Huang M, Zhao J, Huang Y, Dai L, Zhang X. Meta-analysis of urinary C-terminal telopeptide of type II collagen as a biomarker in osteoarthritis diagnosis. J Orthop Translat. 2017 Aug 15;13:50-57. doi: 10.1016/j.jot.2017.06.005. eCollection 2018 Apr. PMID 29662791
- [Background] Hoch JM, Mattacola CG, Medina McKeon JM, Howard JS, Lattermann C. Serum cartilage oligomeric matrix protein (sCOMP) is elevated in patients with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2011 Dec;19(12):1396-404. doi: 10.1016/j.joca.2011.09.005. Epub 2011 Oct 5. PMID 22001901
- [Background] Verma P, Dalal K. Serum cartilage oligomeric matrix protein (COMP) in knee osteoarthritis: a novel diagnostic and prognostic biomarker. J Orthop Res. 2013 Jul;31(7):999-1006. doi: 10.1002/jor.22324. Epub 2013 Feb 19. PMID 23423905
- [Background] Shewale AR, Barnes CL, Fischbach LA, Ounpraseuth ST, Painter JT, Martin BC. Comparison of Low-, Moderate-, and High-Molecular-Weight Hyaluronic Acid Injections in Delaying Time to Knee Surgery. J Arthroplasty. 2017 Oct;32(10):2952-2957.e21. doi: 10.1016/j.arth.2017.04.041. Epub 2017 May 2. PMID 28606459
- [Background] Topol GA, Podesta LA, Reeves KD, Giraldo MM, Johnson LL, Grasso R, Jamin A, Clark T, Rabago D. Chondrogenic Effect of Intra-articular Hypertonic-Dextrose (Prolotherapy) in Severe Knee Osteoarthritis. PM R. 2016 Nov;8(11):1072-1082. doi: 10.1016/j.pmrj.2016.03.008. Epub 2016 Apr 4. PMID 27058744
- [Background] Hung CY, Hsiao MY, Chang KV, Han DS, Wang TG. Comparative effectiveness of dextrose prolotherapy versus control injections and exercise in the management of osteoarthritis pain: a systematic review and meta-analysis. J Pain Res. 2016 Oct 18;9:847-857. doi: 10.2147/JPR.S118669. eCollection 2016. PMID 27799816